CLINICAL TRIAL: NCT03743714
Title: Effects of Yoga Training on Postural Stability and Investigating the Gender-Related Responses
Brief Title: Effects of Yoga Training on Postural Stability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Assoc Prof, Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-292
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Gender; Postural; Defect; Physical Activity
MeSH Terms: conditions — Coitus; Motor Activity | interventions — Pliability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- males (Experimental): healthy, sedentary males
  Interventions: Other: yoga treatment; flexibility, balance and strength exercises.
- females (Experimental): healthy, sedentary females
  Interventions: Other: yoga treatment; flexibility, balance and strength exercises.

INTERVENTIONS:
Other: yoga treatment; flexibility, balance and strength exercises. — yoga treatment including flexibility exercises, balance exercises, and strength exercises.

SUMMARY:
Postural stability can be affected by multiple factors. Such as; body mass, inactivity, age and etc. This study was planned with the aim of investigating the effects of Yoga training on postural stability of males and females. Yoga is a treatment model for body flexibility, body awareness, and strength.

DETAILED DESCRIPTION:
Postural stability can be affected by multiple factors. Such as; body mass, inactivity, age and etc. This study was planned with the aim of investigating the effects of Yoga training on postural stability of males and females. Yoga is a treatment model for body flexibility, body awareness, and strength.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary males and females
* want to participate

Exclusion Criteria:

* have any disorders such as; neurologic, orthopedic, psychiatric or/and systemic.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Sedentary males and females
Enrollment: 24 (Estimated)
Dates: Start 2018-12-02 (Estimated); Primary Completion 2019-11-02 (Estimated); Study Completion 2019-12-02 (Estimated)

PRIMARY OUTCOMES:
Postural stability score | at first minute, at the 2nd day, at the 15th day and at the30th day
  Postural stability score is a composite score including the ability of standing upright position without swing. Individuals stands on a flat platform and perform stepping with possible least changes on their location.

IPD SHARING:
Plan to Share IPD: Undecided